CLINICAL TRIAL: NCT01200875
Title: Effect of Intramuscular and Intratendinous Platelet-Rich Plasma Injections on Systemic Concentrations of Performance-Enhancing Growth Factors
Brief Title: Performance-Enhancing Effects of Platelet-Rich Plasma (PRP) Injections
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Partnership for Clean Competition (Other)
Responsible Party: Principal Investigator, Jason L. Dragoo, Associate Professor, Stanford University
Other Study IDs: SU-08032010-6646; 18963 (Other: Stanford IRB)
Record Dates: First submitted 2010-09-02; First posted 2010-09-14 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Tendinopathy; Rheumatic Diseases
Keywords: PRP; platelet rich plasma; platelet; growth hormone; tendonitis; tendinosis; tendinopathy; enthesopathy; muscle; sport; tendon
MeSH Terms: conditions — Tendinopathy; Rheumatic Diseases; Enthesopathy | interventions — Injections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum, blood plasma, and platelet-rich-plasma (PRP)
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Ultrasound-guided platelet-rich-plasma (PRP) injection — One ultrasound-guided intratendinous or intramuscular PRP injection
Procedure: Platelet-Rich Plasma (PRP) — One ultrasound-guided PRP injection
  Other Names: PRP; Platelet Rich Plasma; Platelet-Rich-Plasma

SUMMARY:
Platelet-Rich Plasma (PRP) has been banned in competitive athletes because some people think it may enhance athletic performance. However, there is very little published research to support or undermine this point of view. The purposes of this study are: (1) To assess the effects of local platelet-rich plasma (PRP) therapy on systemic levels of growth factors with suspected or known performance-enhancing effects; and (2) To understand whether the effect of PRP therapy on these growth factors differs between intramuscular and intratendinous PRP injections.

This research study is looking for 40 people who are receiving platelet-rich plasma therapy for a tendon or muscle injury. The study involves collecting seven blood samples (2 teaspoons each) from each patient, before and after the PRP treatment. Blood samples may be donated at any location of the patient's choosing, and participants will be paid for their time.

DETAILED DESCRIPTION:
To understand the short-term systemic effects of local PRP injections, we will measure the serum concentrations of six growth factors before and during the four days following PRP injection: human growth hormone (hGH), IGF-1, basic FGF, PDGF-BB, VEGF, and IGFBP-3. These molecules are of particular interest because they may have stimulatory effects that enhance athletic performance, and because they have been banned in competitive athletes by the World Anti-Doping Agency (WADA).

We aim to recruit 40 patients who are receiving ultrasound-guided intratendinous (IT) or intramuscular (IM) PRP injections. Blood will be drawn immediately before (baseline); 15 minutes after; and 3, 24, 48, 72 and 96 hours after receiving PRP therapy. A fraction of the therapeutic PRP preparation will be isolated for growth factor analysis. Serum concentrations of growth factors will be quantified by ELISA. Statistical analyses will be conducted to assess the change in each growth factor following PRP injection. To understand the impact of injection site on systemic growth factors, changes in concentration will also be compared between the intratendinous and intramuscular groups.

Study subjects will participate in the following steps: (1) Initial diagnostic visit with Orthopaedic Surgeon, (2) Blood collection as part of PRP therapy, (3) Ultrasound-guided PRP therapy administered by Stanford radiologist, and (4) Blood collection for the study. Steps (1) through (3) are all part of the standard of care, which the patient will have chosen independently of the study. In step (4), blood samples will be collected by venipuncture at various time points and assayed for growth factor concentrations. Less than 10 mL (2 teaspoons) of blood will be collected at each of seven time points over five consecutive days. In order to minimize inconvenience to the patient we will meet patients at a location of their choosing, such as the patient's home or office, for blood collection on days 2-5. Participants will be compensated after all seven blood samples have been donated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18-50 years old, receiving ultrasound-guided intratendinous or intramuscular PRP injections

Exclusion Criteria:

* History of cancer, diabetes, hormone-replacement therapy, or abnormal nutritional habits.
* Contraindications for PRP therapy itself:

  * preexisting coagulation defects including thrombocytopenia
  * hypofibrinogenemia
  * anticoagulation medications
  * hypersensitivity to bovine products, which may be used for platelet activation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving intramuscular or intratendinous platelet-rich-plasma (PRP) for treatment of muscle or tendon injury.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christina Herrero, Study Director — New York University Langone Orthopedic Hospital; Dr. Jason L. Dragoo, Principal Investigator — Stanford University
Locations (1):
- New York University Langone Orthopedic Hospital, New York, New York, United States

REFERENCES:
- [Derived] Wasterlain AS, Braun HJ, Harris AH, Kim HJ, Dragoo JL. The systemic effects of platelet-rich plasma injection. Am J Sports Med. 2013 Jan;41(1):186-93. doi: 10.1177/0363546512466383. Epub 2012 Dec 4. PMID 23211708

RESULTS

PARTICIPANT FLOW:
Groups:
- PRP Injection (All Patients): All patients receiving local ultrasound-guided intratendinous PRP injection at our institution between July 2010 and December 2011 were screened for eligibility to participate in the study, and 25 patients were ultimately enrolled.
Period: Overall Study
Arm/Group | PRP Injection (All Patients)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: All patients receiving local ultrasound-guided intratendinous PRP injection at our institution between July 2010 and December 2011 were screened for eligibility to participate in the study, and 25 patients were ultimately enrolled.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 6
Region of Enrollment [Number; unit: participants] — California, United States
  participants
    United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Blood Growth Factor Concentrations
Time Frame: 5 days following PRP injection
Measure: Mean (95% Confidence Interval); unit: IGF-1 fold-change from baseline @ 24h
Arm/Group | PRP Injection (All Patients)
Number analyzed (Participants) | 25
IGF-1 fold-change from baseline @ 24h | 1.078 [1.009 to 1.148]

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No